CLINICAL TRIAL: NCT01043094
Title: A Study to Compare the Safety, Tolerability, and Pharmacokinetic Profile of a Single Oral Dose of Pitavastatin 4 mg in Adult Volunteers With Severe Renal Impairment Who Are Not Being Treated With Hemodialysis Versus Healthy Adult Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetic of Single Dose of Pitavastatin 4 mg in Severe Renal Patients Versus Healthy Adult Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: NK-104-4.01US
Record Dates: First submitted 2009-12-18; First posted 2010-01-06 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-07

CONDITIONS: Severe Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin 4mg renal impaired (Experimental): Subjects with severe renal impairment (glomerular filtration rate [GFR] of 15 to 29 mL/min/1.73 m2, inclusive) who are not being treated with hemodialysis
  Interventions: Drug: Pitavastatin 4mg
- Pitavastatin 4mg healthy subjects (Active Comparator): Healthy subjects (GFR greater than or equal to 90 mL/min/1.73 m2)
  Interventions: Drug: Pitavastatin 4mg

INTERVENTIONS:
Drug: Pitavastatin 4mg — Pitavastatin 4mg single dose

SUMMARY:
This is a Phase 4, multicenter, open label, 1 period study. A total of 16 subjects are planned (8 subjects in Group A and 8 subjects in Group B):

The 2 groups will be comparable in terms of age, gender, and body mass index (BMI); the ranges for comparison will be obtained from the pooled demographic data of the renally impaired subjects. The mean age of Group B will be within 5 years of the mean age of Group A, the mean BMI of Group B will be within 18% of the mean BMI of Group A, and the ratio of men to women in Group B will be the same as in Group A.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult male or female subject aged 18 years or older. Females of childbearing potential must have a negative pregnancy test before beginning the study.
* Subject has no clinically significant medical conditions (other than renal impairment and associated diseases, such as hypertension, diabetes, and dyslipidemia, for subjects in Group A) as determined by medical history, physical examination, 12-lead ECG, clinical laboratory results (hematology, serum chemistry, and urinalysis [if able to pass urine]), and serology results (hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus types 1 and 2 antibody). Subjects with positive results for hepatitis C virus but who have normal liver enzymes will not be excluded. Any subjects who have impaired hepatic function that will potentially affect drug metabolism should be excluded.
* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is able and willing to comply with the protocol and study procedures.

Exclusion Criteria:

* Subject is on maintenance hemodialysis.
* Subject has a BMI of >37 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period was from 23 November 2009 to 07 June 2010 All subjects were seen at a medical clinic
Period: Overall Study
Arm/Group | Pitavastatin 4mg Renal Impaired | Pitavastatin 4mg Healthy Subjects
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 4mg Renal Impaired | Pitavastatin 4mg Healthy Subjects | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (15.41) | 52.0 (2.62) | 53.1 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0 to Tau (AUC 0-t (ng*h/mL))
Description: Area under the curve from start to elimination for Pitavastatin.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: nanogram hour per milliliter (ng•h/mL)
Arm/Group | Pitavastatin 4mg Renal Impaired | Pitavastatin 4mg Healthy Subjects
Number analyzed (Participants) | 8 | 8
nanogram hour per milliliter (ng•h/mL) | 175 (39) | 145 (55)

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Time Frame: 3 Days
Measure: Number; unit: Participants
Arm/Group | Pitavastatin 4mg Renal Impaired | Pitavastatin 4mg Healthy Subjects
Number analyzed (Participants) | 8 | 8
Participants | 3 | 3

ADVERSE EVENTS:
Arm/Group | Pitavastatin 4mg Renal Impaired | Pitavastatin 4mg Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 4mg Renal Impaired (N=8) | Pitavastatin 4mg Healthy Subjects (N=8)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI not to publish.